CLINICAL TRIAL: NCT05808543
Title: A Randomised Controlled Trial to Evaluate the Effectiveness of Spatial-listening Training Delivered Via the Both EARS Training Package (BEARS) in Older Children and Teenagers With Bilateral Cochlear Implants
Brief Title: BEARS Training Package to Maximise Hearing Abilities in Older Children and Teenagers With Bilateral Cochlear Implants
Acronym: BEARS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: University of Cambridge (Other); University College, London (Other); Imperial College London (Other); University of Nottingham (Other); Cambridge University Hospitals NHS Foundation Trust (Other); University of Southampton (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 319903
Record Dates: First submitted 2023-03-17; First posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-03

CONDITIONS: Hearing Loss, Sensorineural; Hearing Loss; Deafness; Hearing Impaired Children and Adolescents
Keywords: Cochlear Implant; Virtual Reality; Children; Teenagers; Deaf; Bilateral; Training; Rehabilitation
MeSH Terms: conditions — Hearing Loss, Sensorineural; Hearing Loss; Deafness

STUDY DESIGN:
Intervention Model Description: Participants will be randomised on a 1:1 ratio to either the BEARS or usual care intervention arm. The trial will be unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Both EARS training package (BEARS) and Usual Care (Experimental): BEARS is a compilation of virtual reality games designed specifically for young people with bilateral cochlear implants. The hardware is either: A Head Mounted Display Device or an iPad with headphones.
  Interventions: Other: Both EARS training package (BEARS); Other: Usual Care
- Usual Care (Active Comparator): Usual care describes the routine rehabilitation received by participants via their implant centre.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Both EARS training package (BEARS) — The BEARS training package comprises of three games addressing different hearing functions: speech-in-noise perception, music listening and sound-source localisation. Each game is based on an audio-visual task performed through a virtual-reality interface. Players are guided through on-screen visual prompts to support the gameplay with feedback given on their performance and progress through levels of increasing difficulty. The BEARS training package design allows for the training to be self-administered, played anywhere and at any time. There is no upper limit to the frequency of use of the BEARS training package, it is advised to play the games for a minimum of 1 hour a week over a minimum of 2x 30-minute sessions, all three games will need to be played.
  Arms: Both EARS training package (BEARS) and Usual Care
Other: Usual Care — This is an annual review appointment with the patient and their clinician. This could be face-to-face, virtual video consultation, questionnaire, or be cochlear remote care checks. As a minimum this review will check the following: Microphone covers changed, Reported or recorded device use, all external and internal equipment working (known through no reported or recorded degradation in hearing ability). During the appointment, the clinician would establish if there were any concerns regarding the cochlear implant functioning and the patient's rehabilitation programme. They will then make any repairs or adjustments to the device and manage additional support and contact as required. Between the annual review appointments patients can attend the implant centre for repair appointments or have spare equipment posted. There is no limit to the level of contact between the patient and the implant centre.

SUMMARY:
The goal of the BEARS clinical trial is to determine whether using the directional listening training delivered via the BEARS training package for 3-months alongside usual care compared to only receiving usual care improves speech-in-noise perception, hearing experiences, vocabulary and quality of life and reduces listening effort in young people between 8-16 years old (inclusive) with two cochlear implants.

The participants will complete hearing assessments and questionnaires before completing the 3-month intervention. They will be followed up for the next 9-months through online and in-person appointments.

DETAILED DESCRIPTION:
Deafness is the most frequent human sensory deficit. Cochlear implantation is the primary intervention. Currently over 6000 people have bilateral cochlear implants in the United Kingdom, most of these are children.

Two implants are supposed to provide better access to sound, but it is challenging to interpret and integrate what is heard from both sides. Our 'Living with cochlear implants' Patient and Public Involvement group reported that everyday communication is challenging and tiring, with extra effort required to integrate information from two ears, especially in noise. They reported that current rehabilitation techniques are not engaging, or appropriate to their lifestyles.

To address these issues, we have developed a set of virtual reality games called BEARS (Both EARS). BEARS trains sound localisation and listening in noise. These are skills required in everyday listening.

The aim of this trial is to determine whether using the directional listening training delivered via the BEARS training package for 3-months alongside usual care compared to only receiving usual care improves speech-in-noise perception, hearing experiences, vocabulary and quality of life and reduces listening effort in young people between 8-16 years old (inclusive) with two cochlear implants. The study will be carried out in clinical cochlear implant departments in National Health Service or University hospitals.

Participants will be randomly allocated into one of two groups:

1. Receiving the BEARS training package to use for 3-months alongside usual care
2. Continue with usual care

The participants will complete hearing assessments and questionnaires before completing the 3-month intervention. They will be followed up for the next 9-months through online and in-person appointments.

Participants and clinicians can also consent to qualitative or process evaluation interviews, which are BEARS sub-studies

ELIGIBILITY:
Inclusion Criteria:

1. Participant is a simultaneous or sequential bilateral cochlear implant user*, who either has:

   1. Congenital severe/profound bilateral sensorineural hearing loss and have received at least one implant ≤ 36 months of age.
   2. Progressive or acquired severe/profound bilateral sensorineural hearing loss (no age at implant restrictions for these patients) *(a bilateral CI user is defined as a patient who uses both cochlear implant processors for a minimum of 6-hours per day over a month)
2. Participant has stable programmes (defined as no longer using progressive programmes to work through).
3. Participant has had at least two usual care checks/clinical appointments with stable aided levels (+/- 10 dB across 500Hz-4kHz) and no progressive maps to still work through, if they have had re-implantation of internal implant devices.
4. Participant is aged 8-16 years, inclusive.

Exclusion Criteria:

1. Participant (or parent/legal representative) does not speak/understand English sufficiently to undertake assessments.
2. Participant has an intellectual disability at a level that would prevent their ability to understand the trial the intervention or assessment questions.
3. Participant has a comorbid condition impacting ability to participate in the intervention and/or outcome assessment.
4. Participant has an audiological profile impacting ability to participate in the intervention and/or outcome assessments.
5. Participant is actively participating in other trials that may affect hearing outcomes or impact their ability to participate in the intervention.
6. Participant is currently or anticipated to receive treatment and/or intervention that may affect hearing outcomes or adapt implant settings/programming.
7. Participant is refusing to consent to trial activities/protocol.
8. Participant is awaiting reimplantation following device failure or infection.
9. Participant has had any changes to the programmes of either cochlear implant within the last four weeks.
10. Participant has had a change of cochlear implant processor model or upgrade within the last four weeks.
11. Participant is a non-user of one or both implant processors (i.e., must use both processors for a minimum of 6 hours per day over a month).
12. Participant is a fulltime boarder at a boarding school
13. Participant has unresolvable issues found in device checks that render one of the implants unusable.
14. Participant is a female that is pregnant.
15. Participant has a diagnosis of epilepsy or history of seizures of any kind.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 384 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Spatial speech in Noise - Virtual Acoustics (SSiN-VA) test outcome | Three months
  The Primary outcome for the BEARS trial is the difference between the intervention groups in speech-in-noise perception score (% correct overall task) at 3 months, accounting for the participant's baseline score. This is derived from the spatial speech in noise (SSiN-VA) test.

SECONDARY OUTCOMES:
SSiN-VA test outcome | Twelve months
  Speech-in-noise perception score (% correct of the overall task) at twelve months accounting for the baseline score.
SSiN-VA test outcome | Three and Twelve Months
  Relative localisation score (% correct) at three months and at twelve months accounting for the baseline score.
Spatial Adaptive Sentence List (Sp-ASL) test outcomes | Three and Twelve Months
  Speech reception threshold at three months and at twelve months, accounting for baseline (for better ear, worse ear, and average of both).
British Picture Vocabulary Scale (BPVS) test outcome | Twelve Months
  Difference between arms in vocabulary age at twelve months, accounting for baseline vocabulary age
Vanderbilt Fatigue Scale: Child self-report version (VFS-C) questionnaire outcome | Three and Twelve Months
  Difference between arms in listening-related fatigue score at three and 12 months, accounting for baseline.
Speech, Spatial, and Qualities of Hearing Scale for Children with Impaired Hearing (SSQ) outcome | Three and Twelve Months
  Difference between arms in SSQ scores at three and 12 months, accounting for baseline.
Health Economic outcomes | Twelve Months
  The economic evaluation will calculate incremental cost per quality-adjusted life-year (QALY) gained by offering BEARS and usual care, compared to usual care, from an NHS, Personal Social Services (PSS) and Local Education Provider perspective over the twelve months of the trial.
SSiN-VA test outcome | Three and Twelve Months
  Average reaction time (measure of listening effort) for word identification selections at three months and at twelve months accounting for the baseline score.
SSiN-VA test outcome | Three and Twelve Months
  Average reaction time (measure of listening effort) for location shift selection at three months, and at twelve months accounting for the baseline score.
SSiN-VA test outcome | Three and Twelve Months
  Spatial index for word identification at three months and at twelve months accounting for the baseline score.
SSiN-VA test outcome | Three and Twelve Months
  Spatial index for relative localisation at three months and at twelve months accounting for the baseline score.
Spatial Adaptive Sentence List (Sp-ASL) test outcomes | Three and Twelve Months
  Spatial release from masking score at three months and at twelve months, accounting for baseline (for better ear, worse ear, and average of both).

OTHER OUTCOMES:
Age effects | Twelve Months
  No further data will be collected for the age effect analyses but the data regarding the trajectory of the children's speech-in-noise scores relative to normative age range for the speech measures will be assessed to determine if there is a difference in trajectory over time between the BEARS intervention and Usual Care groups.
Retention of training effects | Three and Twelve Months
  No further data will be collected for the retention effect analyses. It is considered best practice in training interventions to evaluate if the training effects remain after the intervention period has finished. For this analysis fixed effects of timepoint (baseline, 3, 6, 9 and 12 months) and group (BEARS intervention, Usual care) and random effect of participant will be used to understand the speech-in-noise outcomes.
Impact of degree of balance between ears | Three and Twelve Months
  For this analysis, the balance app will be used to indicate the degree of symmetry across the two ears. The balance measurements at baseline, three months and 12 months will be used as an outcome to determine if there have been any changes in the balance between the ears over time.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: First year of the trial opening
Access Criteria: Open access

REFERENCES:
- [Result] Vickers D, Salorio-Corbetto M, Driver S, Rocca C, Levtov Y, Sum K, Parmar B, Dritsakis G, Albanell Flores J, Jiang D, Mahon M, Early F, Van Zalk N, Picinali L. Involving Children and Teenagers With Bilateral Cochlear Implants in the Design of the BEARS (Both EARS) Virtual Reality Training Suite Improves Personalization. Front Digit Health. 2021 Nov 12;3:759723. doi: 10.3389/fdgth.2021.759723. eCollection 2021. PMID 34870270
- [Result] Salorio-Corbetto M, Williges B, Lamping W, Picinali L, Vickers D. Evaluating Spatial Hearing Using a Dual-Task Approach in a Virtual-Acoustics Environment. Front Neurosci. 2022 Mar 8;16:787153. doi: 10.3389/fnins.2022.787153. eCollection 2022. PMID 35350560